CLINICAL TRIAL: NCT04376281
Title: The Effect of Norepinephrine on Blood Volume Cardiac , Output and Systemic Filling Pressure in Patients Undergoing Liver Transplant .
Brief Title: The Effect of Norepinephrine on Cardiac Output in Patients Undergoing Liver Transplant .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Hussein Sayed, MD, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD.241-2019
Record Dates: First submitted 2020-04-15; First posted 2020-05-06 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Liver Transplantation
Keywords: Liver transplantaion , fluid management , noradrenaline
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Noradrenaline group (Experimental)
  Interventions: Drug: Noradrenaline

INTERVENTIONS:
Drug: Noradrenaline — Noradrenaline infusion for patients undergoing liver transplantaion from living donor .

SUMMARY:
Early administration of NE in liver transplant recipient might enhance cardiac output through an increase in cardiac preload .

DETAILED DESCRIPTION:
The derangement of circulatory blood volume in patients with liver cirrhosis makes intraoperative fluid management during liver transplant is challenging . Cirrhotic patients not only have large blood volume but abnormal blood volume distribution, with a substantial fraction of this volume in the splanchnic circulation (. These hemodynamic changes render volume loading in these patients has little impact on CO because a large proportion of infused fluid is shifted to the splanchnic system . In addition, patients with liver cirrhosis is similar to septic patients who have increased total vascular compliance which may cause pooling of blood in venous pool. Several studies in patients with sepsis found that use of low dose vasopressor may convert unstressed blood volume (i.e the amount of blood not causing pressure on the vessels) to stressed volume (i.e additional blood causing a distending pressure on the vascular walls and reflects the effective circulating volume) . However, no previous studies tested the effect of using norepinephrine (NE) on venous return and cardiac preload in patients undergoing liver transplant. An obvious advantage of this possibility is that NE will be used instead of true ﬂuid replacement which may minimize fluid replacement during operation.

Recently, a method was described to estimate the changes in intravascular volume and vascular capacitance by calculating mean systemic ﬁlling pressure (MSFP) . MSFP is the driving pressure in venous return, and it allows calculation of the arterial and venous components of systemic vascular resistance .

ELIGIBILITY:
Inclusion Criteria:

* All Adults (age > 18 years) patients undergoing living donor liver transplant (LDLT) will be considered for inclusion in the study..

Exclusion Criteria:

* Patients less than 18 years.
* Patients undergoing liver transplantation for acute liver failure .
* All Chronic Hypertensive patients on medication , whether controlled on not controlled
* Those with high risk of post transplant renal dysfunction (serum creatinine >1.5 mg/dL at time of transplant)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
The effect of Noradrenaline on change of cardiac output . | along the procedure ; from skin incision to the end of surgery
  The effect of Noradrenaline on change of cardiac output .

SECONDARY OUTCOMES:
The effect of NE on mean systemic filling pressure . | along the procedure ; from skin incision to the end of surgery
  The effect of NE on mean systemic filling pressure .
The effect of NE on venous return . | along the procedure ; from skin incision to the end of surgery
  The effect of NE on venous return .
The effect of NE on central venous pressure . | along the procedure ; from skin incision to the end of surgery
  The effect of NE on central venous pressure .

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mukhtar, MD, Study Director — professor
Locations (1):
- kasr El Ainy school of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudnick MR, Marchi LD, Plotkin JS. Hemodynamic monitoring during liver transplantation: A state of the art review. World J Hepatol. 2015 Jun 8;7(10):1302-11. doi: 10.4254/wjh.v7.i10.1302. PMID 26052376
- [Background] Moller S, Bendtsen F, Henriksen JH. Effect of volume expansion on systemic hemodynamics and central and arterial blood volume in cirrhosis. Gastroenterology. 1995 Dec;109(6):1917-25. doi: 10.1016/0016-5085(95)90759-9. PMID 7498657
- [Background] Mukhtar A, Dabbous H. Modulation of splanchnic circulation: Role in perioperative management of liver transplant patients. World J Gastroenterol. 2016 Jan 28;22(4):1582-92. doi: 10.3748/wjg.v22.i4.1582. PMID 26819524
- [Background] Maas JJ, Geerts BF, van den Berg PC, Pinsky MR, Jansen JR. Assessment of venous return curve and mean systemic filling pressure in postoperative cardiac surgery patients. Crit Care Med. 2009 Mar;37(3):912-8. doi: 10.1097/CCM.0b013e3181961481. PMID 19237896